CLINICAL TRIAL: NCT05748405
Title: A Double-blind, Randomized, Placebo-controlled, 4-week, Phase 1/2 Trial in Young Adult Participants With Down Syndrome to Assess the Safety, Tolerability, Plasma Exposure, and Preliminary Indications of Pharmacodynamic Activity of AEF0217
Brief Title: Phase 1/2 Trial of AEF0217 in Participants With Down Syndrome
Acronym: MDDS
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Aelis Farma (Industry)
Collaborators: European Commission (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AEF0217-102; 2022-000923-19 (EudraCT Number)
Record Dates: First submitted 2023-01-11; First posted 2023-02-28 (Actual); Last update posted 2024-10-10 (Actual); Status verified 2024-10

CONDITIONS: Down Syndrome
Keywords: Down Syndrome; Trisomy 21
MeSH Terms: conditions — Down Syndrome

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- AEF0217 (Experimental): AEF0217 0.1 mg tablet 2 tablets in 10 ml of water per day during 28 days
  Interventions: Drug: AEF0217
- Placebo (Placebo Comparator): Placebo tablet 2 tablets in 10 ml of water per day during 28 days
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Placebo — Matching Tablets
  Arms: Placebo
Drug: AEF0217 — Tablets of 100 mcg AEF0217
  Other Names: 3β-benzyloxy-17α-methyl-pregn-5-en-20-one
  Arms: AEF0217

SUMMARY:
AEF0217-102 clinical trial assesses the safety, tolerability, plasma exposure and preliminary indications of pharmacodynamic activity of AEF0217 in female and male adult participants with Down syndrome between 18 and 35 years old.

The trial AEF0217-102 is a double-blind, randomized, placebo-controlled, multiple-dose, 4-week phase 1/2 study. After a screening period, the participant will be randomised and will take an oral dose of AEF0217 0.2mg or placebo once a day for 28 days.

ELIGIBILITY:
Inclusion Criteria:

* Male or female.
* Age ≥18 to ≤35 years.
* Body mass index (BMI) ≥18.5 to ≤32 kg/m2.
* Clinical diagnosis of Down syndrome (full trisomy 21 and translocations) documented by chromosomal analysis (karyotyping).
* Understands and accepts the trial procedures.
* Independently mobile and have sufficient vision and hearing to participate in the trial evaluations.
* Clinical Evaluation of Language Fundamentals Preschool-2 (CELF Preschool-2) test score ≥7.
* IQ >35-70 measured with KBIT. Individuals with IQ from >35 to <40 must have adequate adaptive functioning according to the judgment of the principal investigator.
* Must have a parent or other reliable caregiver who agrees to accompany the participant to all clinic visits and be available for a telephone visit, provide information about the participant as required by the protocol, and ensure compliance with the medication schedule and protocol requirements.
* Vital signs, electrocardiogram (ECG), and safety laboratory parameters must be within normal ranges or without clinically relevant abnormalities except for:

  1. Stable type 1 or type 2 diabetes, i.e., HbA1c level <7%, provided participants are monitored regularly prior to and during the trial to ensure adequate glucose control.
  2. Hypothyroidism provided participants are euthyroid and stable on treatment for at least 6 weeks prior to screening.
* Assent by the participant and consent by the legally authorized representative(s) on behalf of the participant or Consent by the participant in situations where consent rather than assent can be provided by the participant.
* Informed consent by the participant's caregiver to take on the obligations of the caregiver in this trial.

Exclusion Criteria:

* Pregnant or nursing female.
* Mosaic Down syndrome.
* Active or clinically relevant conditions that could, in the investigator's judgment, affect absorption, distribution, or metabolism of the trial intervention (e.g., inflammatory bowel disease, gastric or duodenal ulcers).
* Clinically relevant obstructive pulmonary disease or asthma that is untreated or not controlled by treatment within 6 weeks of screening or being treated with oral steroids.
* Severe obstructive sleep apnea.
* Recent (≤1 year) or ongoing hematologic or oncologic disorders (mild anemia is allowed).
* Personal history of infantile spasms/convulsions/epilepsy, severe head trauma, or CNS infections (e.g., meningitis), except for isolated events of febrile seizures more than 8 years ago.
* Clinically relevant unstable gastrointestinal, renal, hepatic, endocrine, or cardiovascular system disease.
* Current Diagnostic and Statistical Manual of Mental Disorders (DSM-5) diagnosis including autism spectrum disorder or any primary psychiatric diagnosis. Diagnoses that are secondary, such as attention deficit hyperactivity disorder, depression, and conduct disorder are allowed if they are considered not to interfere with the trial conduct and are stable during the 3 months preceding randomization. Medical or behavioral treatments used for stabilization must be on stable regimen and dosing for the last 3 months and the type of treatment must be allowed according to the list of allowed and prohibited medication .
* Treatment with medication known to induce CYP3A4/5 P450 isozymes.
* Intake of vitamin supplements, catechins, or products containing epigallocatechin gallate (EGCG) (e.g., TEAVIGO, Mega Green Tea Capsules Life Extension, or Font-UP Grand Fontaine Laboratories) currently or during the 2 months prior to the baseline assessement.
* Symptoms of early dementia as assessed by the National Task Group-Early Detection Screen for Dementia (NTG-EDSD).
* Disclosure of drug or alcohol abuse during medical interview/anamnesis at screening and/or positive urine test for alcohol or drugs of abuse at screening or/and baseline.
* Epileptiform abnormalities (excluding isolated sharp waves and beyond those expected for age) in the screening EEG performed over 10 minutes with concurrent video recording and evaluated by an expert.
* Participants with a history of suicide attempt or deliberate self-harm due to suicidal ideation. Suicidal ideation (even in the absence of suicide attempt or deliberate self-harm) during the 12 months prior to screening. Assessed by 3 specific questions on suicidal ideation, suicidal behavior, and any self-injurious behavior.
* Known hypersensitivity to any drug.
* Participants with clinically significant illness from 2 weeks prior to screening until Day -1.
* Covid-19 positive test and/or symptoms within the last 10 days prior to Day -1, or according to the requirements of the hospital.
* History of or current life-threatening disease.
* Any other clinically relevant concomitant disease or condition or finding at screening that in the investigator's judgment could jeopardize the participant's safety or interfere with, or the treatment thereof might interfere with, the conduct of the trial and related procedures and/or might bias interpretation of the trial results.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2022-12-15 (Actual); Primary Completion 2024-10-07 (Actual); Study Completion 2024-10-07 (Actual)

PRIMARY OUTCOMES:
Incidence of TEAEs and TESAEs as assessed by ElectroCardioGram (ECG) | Day1, Day 8, Day14, Day21, Day29, Day56
  By evaluating changes from the baseline in ECG parameters
Incidence of TEAEs and TESAEs as assessed by vital signs | Day1, Day4, Day 8, Day14, Day21, Day27, Day 28, Day29, Day42, Day56
  By evaluating changes from the baseline in vital signs
Incidence of TEAEs and TESAEs as assessed by Laboratory clinical parameters | Day1, Day 8, Day14, Day21, Day29, Day56
  By evaluating changes from the baseline in clinical laboratory values from blood and urine samples.
Incidence of TEAEs or TESAEs | From Day1 to Day56
  Assessed by AE and SAE reporting

SECONDARY OUTCOMES:
Potential effects of AEF0217 on cognition using the NIH-ToolBox for ID corrected fluid cognitive | Day1, Day27
  Change from baseline in the corrected fluid cognition composite t-score of the NIH-ToolBox for ID Change from baseline in the scores of each of the individual 5 tests constituting the fluid cognition composite score
Determination of the minimum plasma concentration of AEF0217 before dosing (cthrough) | Day1, Day4, Day8, Day14, Day21, Day22, Day29, Day42, Day56
  AEF0217 concentration will be determined. Ctrough (at steady state) will be estimated based on the plasma concentration-time profile of AEF0217.
Determination of the peak plasma concentration of AEF0217 (Cmax) | Day1, Day4, Day8, Day14, Day21, Day22, Day29, Day42, Day56
  AEF0217 concentration will be determined based on the plasma concentration-time profile of AEF0217 and AEF0217 PK parameter Cmax will be estimated.
Determination of the Time of peak concentration of AEF0217 (Tmax) | Day1, Day4, Day8, Day14, Day21, Day22, Day29, Day42, Day56
  AEF0217 concentration will be determined and AEF0217 PK parameter Tmax will be estimated.
Determination of the plasma half-life of AEF0217 (t1/2) | Day1, Day4, Day8, Day14, Day21, Day22, Day29, Day42, Day56
  AEF0217 concentration will be determined and AEF0217 PK parameter t1/2 will be estimated.
Determination of the Area under the plasma concentration versus time curve of AEF0217 (AUC) | Day1, Day4, Day8, Day14, Day21, Day22, Day29, Day42, Day56
  AEF0217 concentration will be determined, based on the plasma concentration-time profile of AEF0217 and AEF0217 PK parameter AUC will be estimated.
Effect on ElectroEncephaloGram (EEG) parameters | Day28
  Difference between active and placebo at Day 28 in the following EEG parameters:
  * Gamma intertrial coherence (ITC) during an ASSR at 40 Hz.
  * Interhemispheric connectivity (IHC) in resting state (eyes open/closed): Band coherence, phase lag index (PLI).
  * Event-related potential (ERP) associated to novel stimuli in the parietal midline (Pz) during the 3-stimuli oddball task.
  * Cognitive workload and working memory EEG features during the working memory test of CANTAB (Spatial Span Test)

OTHER OUTCOMES:
Responses to treatment according to APOE genotypes. | Day 56
  Determination of the APOE ε4 carriers and non-carriers. Analysis in sub-category
To explore effects on additional ElectroEncephaloGram parameters | Day28
  Difference between active and placebo at Day 28 in the following EEG parameters:
  * Power during an ASSR at 40 Hz.
  * Phase-amplitude coupling and clustering coefficient in resting state (eyes open/closed).

CONTACTS AND LOCATIONS:
Overall Officials: Rafael De la Torre Fornell, Principal Investigator — IMIM
Locations (3):
- Spain (3):
  - Hospital del Mar Medical Research Institute (IMIM),, Barcelona, Catalonia
  - Sant Pau Memory Clinic, Hospital de la Santa Creu i Sant Pau, Barcelona
  - Unidad de Adultos con Síndrome de Down, Hospital de La Princesa, Madrid

REFERENCES:
- See also: The ICOD project, funded by European Union (EU) aims to develop the first pharmacological therapy for cognitive impairment in Down syndrome (DS) making it accessible to patients worldwide. — http://www.icod-project.eu/en/home